CLINICAL TRIAL: NCT00676910
Title: A Phase I Study to Determine the Safety, Pharmacology, and Pharmacodynamics of JNJ26854165 in Subjects With Advanced Stage and/or Refractory Solid Tumors
Brief Title: A Research Study of JNJ-26854165 to Determine the Safety and Dose in Patients With Advanced Stage or Refractory Solid Tumors.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR012745
Record Dates: First submitted 2008-05-08; First posted 2008-05-13 (Estimated); Last update posted 2010-03-26 (Estimated); Status verified 2010-03

CONDITIONS: Neoplasms
Keywords: Advanced Cancer; Malignancies; Neoplasms; Incurable Solid Cancers
MeSH Terms: conditions — Neoplasms | interventions — JNJ 26854165

INTERVENTIONS:
Drug: JNJ-26854165

SUMMARY:
The purpose of this study is to assess the safety of JNJ-26854165 (a new drug in development for cancer) in patients with advanced or refractory solid tumors on the maximum dose tolerated by these patients.

DETAILED DESCRIPTION:
JNJ-26854165 is a new drug in development and belongs to a class of drugs that act on the specific protein present in cells. It may stop cancer cells from growing or kill cancer cells. In this study, the safety (the effect on the body) of the JNJ-26854165 in patients with advanced or refractory solid tumors will be examined. The effect (if any) of JNJ-26854165 on the disease will be assessed throughout the study. The maximum dose tolerated by these patients will be determined.

The dose of JNJ 26854165 will start low and will be increased during the study. The drug will be taken by mouth every day in each 21-day cycle. The dose each patient receives will be assigned at enrollment. Patients who enroll at a later time may receive a higher dose. If patients do not have severe side effects at a certain dose level, the next group of 3 to 6 patients will get a higher dose. The dose will increase until some patients have severe side effects. The dose will be then decreased and 3 to 6 patients will receive the highest amount of drug where non-severe side effects were observed.

The amount of JNJ 26854165 in the blood will be measured and the effect of JNJ 26854165 on the disease will also be monitored. The effect of food on the absorption, break down and elimination of the drug will be studied in some patients. At some dose levels, the possible interaction of JNJ 26854165 with medications frequently used in cancer patients will be examined and patients at these dose levels will be asked to take a single dose of three additional drugs (dextromethorphan hydrobromide (30mg), tolbutamide (250mg), and midazolam (5mg) "cocktail") on 2 study days, which will all be supplied by the study doctor.

Patients will be screened for eligibility up to 4 weeks before the study drug is administered. During Cycle 1 patients will be observed as inpatients for at least 12 hours after administration of the drug on 3 or 4 days and will be required to visit the study site on 2 additional days. One additional visit is required for patients in whom the food effect or interaction with other medications will be examined. During Cycle 2, patients are required to visit the study center on 2 days. During all cycles after Cycle 2, patients are required to visit the study center on 1 day. Fourteen days after the last dose of JNJ-26854165, the patient will be invited for a follow-up visit which will include tests for safety and the effect of the drug on the disease. The proposed starting dose of JNJ-26854165 is 4 mg/day as a single oral dose. JNJ26854165 will be provided in a glass vial with tear-off cap placed in a child resistant pouch so that the drug may be taken at home. Patients will take JNJ-26854165 each day while in the study. Treatment may continue as long as there is benefit and there are no unacceptable side effects as assessed by the study doctor.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed solid malignancy, in advanced, incurable stage or not responsive to available therapies
* performance status (based on the Eastern Cooperative Oncology Group assessments) of <= 2
* life expectancy > 3 months
* must consent to skin biopsies
* must meet protocol-defined criteria for lab assessments and heart function.

Exclusion Criteria:

* Known central nervous system metastasis
* chemotherapy, radiotherapy, immunotherapy or use of any investigational agent within 2 weeks before dosing
* treatment within last 6 months or expected to require treatment with amiodarone derivates during study participation
* currently treated and/or expected to require treatment with warfarin/coumarine derivates during study participation
* history of uncontrolled heart disease or uncontrolled arterial hypertension
* eye abnormality at screening examination
* >70% stenosis of lumen on Carotid duplex assessment at screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2006-11; Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Determine the safety of JNJ-26854165 and the maximum tolerated dose in patients with advanced stage or refractory solid tumors.

SECONDARY OUTCOMES:
Determine how JNJ-26854165 is absorbed, broken down and eliminated and the effect of food on these processes. Explore how JNJ-26854165 effects the body and the disease.Determine how JNJ-26854165 interacts with other specific drugs.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.